CLINICAL TRIAL: NCT02388477
Title: Randomized Controlled Trial of the Use of Doxycycline After Rotator Cuff Repair
Brief Title: Trial of the Use of Doxycycline After Rotator Cuff Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research idea tabled at this point.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Aman Dhawan, MD, Assistant Professor of Surgery, Orthopaedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002143
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Rotator Cuff Injury
Keywords: rotator cuff repair; Doxycycline
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Doxycycline; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Active Comparator): oral doxycycline, 2 weeks, twice a day,
  Interventions: Drug: Doxycycline
- sugar pill (Placebo Comparator): sugar pill, same size, shape, and color as comparator, twice a day for 2 weeks.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Doxycycline — antibiotic used to treat infection
  Other Names: Oracea,; Doryx; Monodox; Vibra-Tabs; Morgidox; Periostat; Atridox; Ocudox; Alodox
  Arms: Doxycycline
Drug: sugar pill — placebo with no pharmacologic effect
  Arms: sugar pill

SUMMARY:
The purpose of this study is to examine healing after rotator cuff repair in subjects either treated with Doxycycline or placebo post-operatively.

DETAILED DESCRIPTION:
Basic Science small animal model data indicates that matrix metalloproteinase (MMP) inhibition via doxycycline results in improved early rotator cuff repair biomechanics and histology. Rotator cuff repair failure and retear is a significant clinical problem. The effects of MMP inhibition on human rotator cuff tear repair healing and outcomes is unknown, but may potentially improve healing rates and outcomes. Our purpose is to evaluate the effects of early oral doxycycline on healing and outcomes following arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* repair of rotator cuff
* age 18 and above
* able to swallow capsules

Exclusion Criteria:

* less than 18
* unable to read or understand consent form
* unable to swallow capsules
* allergy to doxycycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
rotator cuff ultrasound of post-operative shoulder | one year
  An ultrasound of the post-operative rotator cuff to assess level of healing or defect present.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons score | 6 weeks, 3mos, 6mos, 1yr and 2 yr.
  The survey is a standardized assessment of shoulder pain and function from the patient's perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Aman Dhawan, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States